CLINICAL TRIAL: NCT06339190
Title: A Blood Test for Dementia? A Cohort Study to Assess the Diagnostic Utility of Plasma Neurofilament Light Chain Protein in All-cause Dementia
Brief Title: Neurofilament Light Chain And Voice Acoustic Analyses In Dementia Diagnosis
Acronym: NAVAIDD
Status: Recruiting | Type: Observational
Sponsor: Monash University (Other)
Collaborators: Eastern Health (Other); University of Melbourne (Other); Wake Forest University (Other); Deakin University (Other); The Florey Institute of Neuroscience and Mental Health (Other); Invitae Corporation (Industry); Redenlab (Unknown)
Responsible Party: Principal Investigator, Amy Brodtmann, Professor, Monash University
Other Study IDs: E21-006-72840
Record Dates: First submitted 2023-09-21; First posted 2024-04-01 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Neurodegenerative Diseases; Dementia
Keywords: Alzheimer's disease; Dementia; Neurofilament light chain; Speech; Neurodegeneration; Biomarker; Health care disparity
MeSH Terms: conditions — Neurodegenerative Diseases; Dementia; Alzheimer Disease; Charcot-Marie-Tooth disease, Type 1F; Speech; Nerve Degeneration | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be used and processed for plasma and Nfl levels will be quantified using the Quanterix HD-X machine and single molecule array (Simoa).
  All participants will be offered participation in DNA and plasma banking for future research as an optional part of the study. DNA samples from participants who consent to this optional collection of plasma will contribute to international biobanking initiatives.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Venepuncture — A single blood draw at the time of presentation to clinic or whilst an inpatient.

SUMMARY:
This cohort study aims to determine if a blood test can aid with diagnosing dementia in anyone presenting with cognitive complaints to a single healthcare network. The investigators will measure levels of a brain protein, Neurofilament light chain (Nfl), and assess changes in language using speech tests.

Participants will have a single blood test and speech test, and will be followed up at 12-months to complete questionnaires and cognitive scales over the phone. The speech test will also be completed again at 12-months.

Individuals at risk of a Fronto-temporal dementia syndrome will be eligible to complete optional genetic testing involving an 'at home' saliva sample.

DETAILED DESCRIPTION:
Problem: There is no "gold-standard test" to detect all forms of dementia. People can present with subtle changes that are missed on standard cognitive screening tests, which are not designed for people whose first language is not English or from diverse cultural and educational backgrounds. State-of-the art brain imaging is only available to Australians living in large urban centres, further entrenching health care inequities. The lack of validated diagnostic tests and pathways causes diagnostic delays, increases patient and caregiver stress. Therapies are on the horizon for many forms of dementia - not only Alzheimer's disease - meaning that the lack of identification of simple dementia diagnostic biomarkers represents a critical knowledge gap.

Mission: New technologies now allow us to test abnormal brain protein levels in a routine peripheral blood test, record a voice sample to analyse its acoustics and reveal brain disease, and perform "mail-out" genetic tests using a simple saliva sample. The levels of a brain derived blood protein, neurofilament light chain (NfL), will be estimated and natural language processing and acoustic analysis will be measured in all patients presenting with cognitive complaints to a single healthcare network servicing 1 million ethnically and culturally diverse Australians. Researchers will investigate the utility of early genetic testing for those at high risk of a genetic cause for their disease. They will use these data to develop diagnostic pathways, leveraging existing collaborations to develop future screening programs. Early to mid-career researchers will be supported to translate new technologies into clinical practice in the shortest practicable time-frame.

Significance: Accessible and cost effective tests will inform new pathways to dementia diagnosis. This will transform the dementia landscape, shortening time to diagnosis, increasing diagnostic certainty, and allowing more Australians access to appropriate care, education, and future therapies.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to Eastern Health services with a cognitive complaint or potential neurodegenerative disorder

Exclusion Criteria:

* Prognosis <12 months
* No cognitive complaint
* Patients not involved within the single healthcare network

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study cohort will include any individual of all ages, ethnicities, identities and genders. This is to ensure that the findings are generalisable to other national healthcare networks and to provide maximum information on the utility of using blood-biomarker estimation in real-world clinical settings
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Baseline NfL level | Day 0
  Plasma Nfl (pg/ml), estimated using Quanterix SIMOA HD-X

SECONDARY OUTCOMES:
Change in speech processing | Day 0 and 12-months
  Staff and/or self administered using Redenlab software and analysed by speech pathologist for acoustic measures of timing (e.g., pause length (seconds) in reading and monologue tasks), vocal control (e.g., fundamental frequency (hertz) and loudness variation (decibel) from vowel and monologue), and vocal quality (e.g., dysphonia measures derived from sustained vowel).
Change in language processing | Day 0 and at 12-months
  Recorded by a member of the research team using Redenlab software and assessed by a speech therapist using Natural Language Processing techniques.
Change in Direct Magnitude Estimation | Day 0 and at 12-months
  Perceptual rating of speech using Redenlab software; measuring intelligibility (i.e ability to be understood) and naturalness (deviation from healthy norm) of speech. Assessed by a speech therapist on a scale from 0 to 100; 0 indicates none of the speech is intelligible/natural, 100 indicates all the speech is intelligible/natural.

OTHER OUTCOMES:
Modified Rankin Scale | Day 0 and at 12-months
  Functional screen; assessed by member of the research team based on clinical notes. Assessed as change from baseline. Scores ranging from 0-5, with higher scores indicating greater disability.
Montreal Cognitive Assessment score | At 12-months
  Cognitive screen; staff administered via telephone. Scores include overall MoCA score (0-22) and Memory Index Score (0-15), greater scores indicate greater cognition.
Hospital Anxiety and Depression Scale score | At 12-months
  Mood screen; staff administered via telephone. Scores include a total depression score (0-21) and total anxiety score (0-21); grouped according to normal (0-7), Borderline abnormal (8-10) and Abnormal (11-21).
Clinical Global Impression score | At 12-months
  Global rating of improvement/change; staff administered via telephone. Scored on a 7 point scale, scores closer to 0 indicative of greater improvement and scores closer to 7 representing much worse).
WHO Disability Assessment 12-item telephone interview score | At 12-months
  Functional screen, staff administered via telephone. Scored as an overall percentage (%) disability, higher scores indicating less function.
WHO Disability Assessment 36-item self report score | At 12-months
  Functional screen, self administered. Scored as an overall percentage (%) disability, higher scores indicating less function.
DNA sample for testing known pathogenic dementia mutations | Anytime before 12-months
  Self-administered saliva sample; Testing using Invitae Fronto-temporal dementia and AD panel: C9orf72, CHCHD10, CHMP2B, DCTN1, FUS, GRN, HNRNPA2B1, MAPT, SQSTM1, TARDBP, TBK1, TREM2, UBQLN2, VCP

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Amy Brodtmann, MBBS, FRACP, PhD, FANZAN, Principal Investigator — Monash University
Locations (2):
- Australia (2):
  - Box Hill Hospital, Box Hill, Victoria
  - Wantirna Health, Wantirna, Victoria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ivanic S, Vogel AP, Chatterjee P, Baird J, Darby D, Werden E, Gao L, Darzins P, Patel SK, Burke I, Morris T, Churilov L, Bice J, Mielke MM, Brodtmann A. Neurofilament light chain and voice acoustics in dementia diagnosis (NAVAIDD): Protocol for a cohort study assessing the real-world diagnostic utility of blood and digital biomarkers in clinical settings. J Alzheimers Dis Rep. 2025 Dec 15;9:25424823251395325. doi: 10.1177/25424823251395325. eCollection 2025 Jan-Dec. PMID 41409494

DOCUMENTS (1):
  • Informed Consent Form (2025-03-11): https://cdn.clinicaltrials.gov/large-docs/90/NCT06339190/ICF_000.pdf